CLINICAL TRIAL: NCT04013932
Title: Family Psychoeducation for Adults With Psychotic Disorders in Tanzania (Pilot Clinical Trial of KUPAA)
Brief Title: Family Psychoeducation for Adults With Psychotic Disorders in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00094163; 5R34MH106663 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders, Severe
Keywords: Family Psychoeducation; Schizophrenia; Tanzania; Severe and Persistent Mental Illness; Culturally tailored
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders; Schizophrenia

STUDY DESIGN:
Masking Description: Only the main biostatistician will be masked in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KUPAA Intervention + Standard of Care (Experimental): Patients will be assigned to a KUPAA group composed of approximately 6 patients (joined by their 6 matched caregivers). Patients will first participate in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop. Participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks.
  Interventions: Behavioral: KUPAA Intervention Group (Culturally Tailored Family Psychoeducation)
- Control - Standard of Care (No Intervention): Patients will receive the standard of care.

INTERVENTIONS:
Behavioral: KUPAA Intervention Group (Culturally Tailored Family Psychoeducation) — KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
  Other Names: FPE; Family psychoeducation
  Arms: KUPAA Intervention + Standard of Care

SUMMARY:
The goal of this study is to pilot test a culturally tailored Family Psychoeducation model (KUPAA) for adults with psychotic disorders and their relatives that is appropriate for cultural settings inclusive of both traditional and biomedical ideas about mental illness and that incorporates relatives as co-facilitators of the intervention.

DETAILED DESCRIPTION:
Family psychoeducation (FPE) is an evidence-based practice used in high-income countries to help individuals with psychotic disorders and their relatives to cope more effectively with the illness. FPE has never been tested in a low-resource country nor have the mechanisms of action for this psychosocial intervention been fully identified in any context. The goal of this study is to pilot test a culturally tailored Family Psychoeducation model (called KUPAA) for adults with psychotic disorders and their relatives that is appropriate for cultural settings inclusive of both traditional and biomedical ideas about mental illness and that incorporates relatives as co-facilitators of the intervention. Formative research has already been conducted to culturally tailor the model for the Tanzanian context. This pilot study is a small randomized controlled trial (RCT) with 72 patient/relative dyads that will test the KUPAA intervention to a) assess the feasibility and acceptability of the adapted family psychoeducation intervention for 12 weeks, and b) explore its impact on patient relapse, quality of life and disability.

Primary study objectives

1. To pilot test the KUPAA intervention to explore its impact on patient relapse, quality of life and disability

   Secondary study objectives
2. To elucidate the mechanisms of action for KUPAA (e.g. hopefulness, self-efficacy) and refine the mediation and study outcome measures for a future R01/fully powered clinical trial

ELIGIBILITY:
Patient Inclusion Criteria:

* Attending outpatient psychiatric services at Muhimbili National Hospital (MNH) or Mbeya Zonal Referral Hospital (MZRH).
* ICD-10 Diagnosis of a non-organic psychotic disorder:
* F20 Schizophrenia
* F21 Schizotypal disorder
* F22 Delusional disorders
* F25 Schizoaffective disorders
* Age 18-50 at the time of informed consent
* Hospitalization or relapse (confirmed by attending psychiatrist or medical officer) within the past 12 months.

Patient Exclusion Criteria:

* F23 Brief psychotic disorder
* F28 Other psychotic disorder not due to a substance or known physiological condition
* F29 Unspecified psychosis not due to a substance or known physiological condition
* Epileptic psychoses
* Bipolar disorder and mania
* Co-morbid developmental disorder, dementia, or other severe cognitive deficit that renders the individual unable to provided informed consent.

Caregiver Inclusion Criteria:

* Age 18 or older at time of consenting process
* Patient agrees that this person can be their paired partner for KUPAA if the pair is randomized to the intervention group

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy Noel Baumgartner, PhD, Principal Investigator — Duke University
Locations (2):
- Tanzania (2):
  - Muhimbili University of Health and Allied Sciences (MUHAS), Dar es Salaam
  - Mbeya Zonal Referral Hospital, Mbeya

IPD SHARING:
Plan to Share IPD: Yes
Adhering to NIMH requirements on sharing data through NIMH Data Archive
Supporting Information: Study Protocol, SAP
Time Frame: By November, 2020
Access Criteria: NIMH Data Archive
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Egger JR, Kaaya S, Swai P, Lawala P, Ndelwa L, Temu J, Bukuku ES, Lukens E, Susser E, Dixon L, Minja A, Clari R, Martinez A, Headley J, Baumgartner JN. Functioning and quality of life among treatment-engaged adults with psychotic disorders in urban Tanzania: Baseline results from the KUPAA clinical trial. PLoS One. 2024 Jun 18;19(6):e0304367. doi: 10.1371/journal.pone.0304367. eCollection 2024. PMID 38889160
- [Derived] Martinez A, Baumgartner JN, Kaaya S, Swai P, Lawala PS, Thedai B, Minja A, Headley J, Egger JR. Hopefulness among individuals living with schizophrenia and their caregivers in Tanzania: an actor-partner interdependence model. BMC Psychiatry. 2023 Jul 13;23(1):508. doi: 10.1186/s12888-023-04990-8. PMID 37442999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At enrollment, all patients had to identify a caregiver for study participation. If the patient was randomized to the intervention arm, the caregiver would participate in the KUPAA groups with the patients. If the patient was randomized to the control arm, there was no interaction with the caregiver beyond standard of care. All data are focused on the patients only for primary outcomes as they are primary unit of analysis.
Groups:
- KUPAA Intervention + Standard of Care: Patients will be assigned to a KUPAA group composed of approximately 6 patients who will also be joined by their caregivers in their sessions. The patients will first participate in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop open to both the patients and their caregivers. Patient-participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks with their caregiver.
  KUPAA Intervention Group (Culturally Tailored Family Psychoeducation): KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
Period: Overall Study
Arm/Group | KUPAA Intervention + Standard of Care | Control - Standard of Care
Started | 33 | 33
Completed | 33 | 28
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Population: The primary analysis population is the patients and that is what is reported in the tables (not caregivers). Patients could participate in the intervention arm even if a caregiver stopped attending group sessions. The intervention is focused on patient outcomes (disability, quality of life, and relapse).
Groups:
- KUPAA Intervention + Standard of Care: Patients will be assigned to a KUPAA group composed of approximately 6 patients and 6 matched caregivers. The dyads will first participate in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop. Participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks.
  KUPAA Intervention Group (Culturally Tailored Family Psychoeducation): KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
- Total: Total of all reporting groups
Arm/Group | KUPAA Intervention + Standard of Care | Control - Standard of Care | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.64 (8.52) | 32.45 (7.94) | 33.05 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 20 | 24 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of participants in Tanzania
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 33 | 33 | 66
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 33 | 33 | 66
4 or more years since illness onset [Count of Participants; unit: Participants] | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patient Participants Who Experience Illness Relapse
Description: Patient relapse measured by hospitalization or non-hospitalized relapse, defined as a new illness episode with recurrence of symptoms after one month of controlled symptoms.
Time Frame: Relapse is measured from immediate post-intervention to endline (~6-7 months post-intervention)
Population: Data not collected on two Control participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- KUPAA Intervention + Standard of Care: Patients will be assigned to a KUPAA group composed of approximately 6 patients (who attend with a matched caregiver). Participants first participate in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop. Participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks.
  KUPAA Intervention Group (Culturally Tailored Family Psychoeducation): KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
Arm/Group | KUPAA Intervention + Standard of Care | Control - Standard of Care
Number analyzed (Participants) | 33 | 31
proportion of participants | 0.27 [0.13 to 0.46] | 0.45 [0.27 to 0.64]

2. Primary Outcome: Change From Baseline to Endline in Disability, as Measured by the World Health Organization Disability Assessment Schedule Version 2.0 (WHODAS 2.0)
Description: Scores are measured from the 36-item WHODAS 2.0, the World Health Organization Disability Assessment Schedule, which measures health and disability. WHODAS 2.0 This self-report assessment measures difficulties performing daily activities over the past 30 days. It consists of 36 Likert-formatted questions across six domains: understanding and communicating, getting around, self-care, getting along with others, life activities, and participation in society. WHO's guidelines for the complex scoring method were used to create the total score, ranging from 0 (no disability) to 100 (full disability). Higher scores indicate worse outcomes.
Time Frame: Baseline (pre-intervention) and Endline (~6-7 months post-intervention)
Population: Data not collected on five Control participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- KUPAA Intervention + Standard of Care: Patients will be assigned to a KUPAA group composed of approximately 6 patients (with their matched caregivers). Patients participated in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop. Participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks.
  KUPAA Intervention Group (Culturally Tailored Family Psychoeducation): KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
Arm/Group | KUPAA Intervention + Standard of Care | Control - Standard of Care
Number analyzed (Participants) | 33 | 28
units on a scale | 14.89 (14.66) | 26.67 (21.58)

3. Primary Outcome: Change From Baseline to Endline in Quality of Life, as Measured by the World Health Organization Quality of Life- Abbreviated Version (WHOQOL-BREF)
Description: Raw total scores are measured from the 26-item WHOQOL-BREF (the abbreviated version of the World Health Organization Quality of Life 100 scale). This self-report assessment has 26 questions across four domains; physical health, psychological, social relationships, and environment. Each item is rated on a five-point Likert scale (1-5) ranging from 1 (not at all, very dissatisfied, very poor) to 5 (an extreme amount, very satisfied, very good); three items needed reverse scoring. The range is 26 (min) to 130 (max) for the total raw score. Higher scores indicate a better outcome.
Time Frame: Baseline (pre-intervention) and Endline (~6-7 months post-intervention)
Population: Data not collected on five Control participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- KUPAA Intervention + Standard of Care: Patients will be assigned to a KUPAA group composed of approximately 6 patients (with their matched caregivers). Patients will first participate in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop. Participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks.
  KUPAA Intervention Group (Culturally Tailored Family Psychoeducation): KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
Arm/Group | KUPAA Intervention + Standard of Care | Control - Standard of Care
Number analyzed (Participants) | 33 | 28
units on a scale | 94.88 (20.98) | 77.39 (16.95)

ADVERSE EVENTS:
Time Frame: From baseline to endline data collection (~1 year)
Description: Adverse event data was not collected on caregivers. Death and temporary missing person experiences were identified during follow-up data collection timepoints (review of medical records and contacts with caregivers).
Groups:
- KUPAA Intervention + Standard of Care: Patients will be assigned to a KUPAA group composed of approximately 6 patients per group (with matched caregivers also attending). Patients first participate in 1-2 joining sessions with a provider, followed by a 1-day group educational workshop. Participants will then attend weekly family psychoeducation group sessions (~1.5-2 hours) for 12 weeks.
  KUPAA Intervention Group (Culturally Tailored Family Psychoeducation): KUPAA is composed of 3 key components:
  1-2 Joining sessions [~30 to 45 minutes each] give the facilitator and participants a chance to get to know each other before KUPAA groups begin and allows time for questions.
  Educational Workshop is an interactive, one day workshop offering information about biological, psychological and social aspects of mental illness; the nature, effects and side effects of psychiatric treatments; what families can do to help recovery and prevent relapse; and guidelines for managing mental illnesses.
  12 Family psychoeducation group sessions [~1.5 hours each session] occur weekly in multi-family groups. These sessions follow an empirically tested format and focus on solving problems that interfere with treatment, illness, and symptoms management and that support coping skills and personal care. Case management may also be provided.
Arm/Group | KUPAA Intervention + Standard of Care | Control - Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/33 | 1/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 2/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KUPAA Intervention + Standard of Care (N=33) | Control - Standard of Care (N=33)
Patient who left home temporarily/missing (relapse related) (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT04013932/Prot_SAP_002.pdf